CLINICAL TRIAL: NCT00477347
Title: Comparison of Manual Propofol and Remifentanil Administration and Dual Closed-loop, Using Bispectral Index as the Control Variable, During Liver Transplantation
Brief Title: Closed-loop Anesthesia, Using Bispectral Index as the Control Variable, During Liver Transplantation
Acronym: Drone-TH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recrutment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006/37
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Anesthesia, general; Closed-loop

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Manual administration
  Interventions: Device: Manual administration
- 2 (Experimental): Closed-loop administration
  Interventions: Device: Closed loop administration

INTERVENTIONS:
Device: Closed loop administration — intraoperative closed loop administration of propofol and remifentanil
  Other Names: closed-loop
  Arms: 2
Device: Manual administration — intraoperative manual administration of propofol and remifentanil
  Other Names: target controlled anesthesia
  Arms: 1

SUMMARY:
To compare closed-loop anesthesia to manual administration of propofol and remifentanil during liver transplantation

DETAILED DESCRIPTION:
The Bispectral Index (BIS) is an electroencephalogram-derived measure of anesthetic depth. We hypothesized that BIS can also indicate the adequacy of analgesia. Therefore we built a combined closed-loop anesthesia system using BIS as control variable and two proportional-differential control algorithms, a propofol and a remifentanil target-controlled infusion system. The effectiveness of such a closed-loop anesthesia system has been demonstrated in a prospective, randomized study.

Elimination of anesthetic agents, propofol in particular, is strongly reduced during liver transplantation. Closed-loop anesthesia could provide adequacy for requirements in respect to the various phases of transplantation. Two groups of patients are compared: one in which propofol and remifentanil are administered by the anesthesiologist, using target-controlled infusion systems, and one in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups the goal is to maintain BIS between 40 and 60, the range recommended by the manufacturer during anesthesia. We expect the combined closed-loop anesthesia system group to do better: i.e. diminished consumption of propofol (primary outcome measure).

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation

Exclusion Criteria:

* pregnant women
* allergy to propofol or remifentanil,
* neurological or muscular disorder,
* liver encephalopathy,
* patients taking psychotropic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
consumption of propofol during anesthesia maintenance | during anesthesia maintenance

SECONDARY OUTCOMES:
- consumption of remifentanil - target modifications - hemodynamic events - volume loading and transfusion - extubation time, explicit memorization - time passed at BIS between 40 and 60 - MDAPE, wobble - global score - dysfunction of each system. | during anesthesia maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Principal Investigator
Locations (2):
- France (2):
  - Dept of Anesthesia and Intensive Care, Hôpital Beaujon, Clichy
  - Dept of Anesthesia and Intensive Care, Hôpital H. Mondor, Créteil

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963